CLINICAL TRIAL: NCT05972343
Title: COOL-IT-PRO: Cryoablation of Breast Cancer in Non-surgical Patients: A Prospective Observational Registry
Brief Title: COOL-IT-PRO: Cryoablation of Breast Cancer in Non-surgical Patients
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 202307067
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cryoablation: Following pre-procedural imaging evaluation, patients will receive ultrasound-guided percutaneous cryoablation as part of their routine treatment of their breast cancer. Follow up imaging (if tolerated) will be performed at 6 months and 12 months and annually thereafter for until 3 years post-procedure. Data will be collected on patient demographics, disease characteristics, treatment, treatment complications, follow-up imaging, response (for 3 years post-procedure), and quality of life.
  Interventions: Device: Cryoablation

INTERVENTIONS:
Device: Cryoablation — Takes place at single time point.

SUMMARY:
This is a subject registry study of patients who undergo cryoablation for their breast cancer after being determined not to be surgical candidates. Data collected as part of this registry will be used to assess the safety of percutaneous ultrasound-guided cryoablation in this population as well as provide long-term follow-up of subjects who received cryoablation.

ELIGIBILITY:
Eligibility Criteria:

* Diagnosis of breast cancer.
* Mass must be visible on ultrasound and > 5 mm from skin.
* Not undergoing surgery, because:

  * Patient has a medical condition that would not allow sedation or general anesthesia
  * Surgery is not clinically indicated due to unresectable and/or metastatic disease
  * Surgery is not clinically indicated for another reason
  * Patient declines surgery
* At least 18 years old.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at Siteman Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2031-07-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who are free of serious treatment related complications per CTCAE v 5.0 | Through 3 year follow-up

SECONDARY OUTCOMES:
Proportion of patients who demonstrate progression-free survival (PFS) | At 3 year follow-up
Proportion of patients who demonstrate disease-free survival (DFS) | At 3 year follow-up
Proportion of patients who demonstrate overall survival (OS) | At 3 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Heather Garrett, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
In addition to the analyses proposed in this protocol, the data collected under this registry will be stored for potential (currently unknown) research projects and may be used to query for feasibility of future projects and other quality initiatives.
Supporting Information: Study Protocol, SAP
Access Criteria: Requests from individuals outside Washington University will require a formal data use agreement (DUA) before release of data for limited data sets and/or identifiable data sets.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu